CLINICAL TRIAL: NCT01810939
Title: A Two-Part, Single-Blind, Phase 3 Study Evaluating the Efficacy and Safety of Patiromer for the Treatment of Hyperkalemia
Brief Title: A Two-Part, Single-Blind, Phase 3 Study Evaluating the Efficacy and Safety of Patiromer for the Treatment of Hyperkalemia (OPAL)
Acronym: OPAL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Relypsa, Inc. (Industry)
Responsible Party: Sponsor
Organization: Vifor Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RLY5016-301; 2012-001956-20 (EudraCT Number)
Record Dates: First submitted 2013-03-12; First posted 2013-03-14 (Estimated); Results first posted 2015-12-15 (Estimated); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: Chronic Kidney Disease (CKD); Hyperkalemia (HK)
Keywords: Chronic Kidney Disease; Treatment of Hyperkalemia; Hyperkalemia
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperkalemia | interventions — patiromer; Suspensions

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patiromer (Active Comparator): Patiromer was administered twice a day as a powder mixed with water.
  Interventions: Drug: Patiromer
- Placebo (Placebo Comparator): Placebo was administered twice a day as a powder mixed with water.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Patiromer
  Other Names: RLY5016 for Oral Suspension; Veltassa
  Arms: Patiromer
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study was to evaluate the efficacy and safety of patiromer (investigational drug) in the treatment of hyperkalemia (high serum potassium). The study also evaluated the effect of withdrawing patiromer treatment and assessed whether chronic treatment with patiromer prevented the recurrence of hyperkalemia. The safety of patiromer treatment was also evaluated.

DETAILED DESCRIPTION:
There were two parts in the study, Part A and Part B.

Part A was an assessment of 4 weeks of dosing with patiromer in the treatment of hyperkalemia; Part B was a randomized, placebo-controlled, 8-week assessment of the withdrawal of patiromer in participants with a baseline serum potassium at the beginning of Part A ≥ 5.5 mEq/L who responded to the 4 weeks of treatment with patiromer during Part A.

All participants received patiromer during Part A; Part B participants were randomized to continue patiromer or switch to placebo. Total study participation was up to 14 weeks (including up to 2 weeks of follow up).

The dose of patiromer could be titrated based on participant's serum potassium response.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ages 18 - 80
* Chronic kidney disease (CKD) - eGFR 15 to < 60 mL/min/1.73m2 at screening
* Hyperkalemia, defined as a serum potassium value of 5.1 to < 6.5 mEq/L at screening
* Taking either an Angiotensin-Converting Enzyme (ACE) Inhibitor, an Angiotensin II receptor blocker (ARB), or an aldosterone antagonist (AA) medication
* Informed consent given

Exclusion Criteria:

* Participants with auto-immune related chronic kidney disease such as lupus nephritis or renal scleroderma/scleroderma renal crisis, or mixed connective tissue disease with renal involvement
* Participants with uncontrolled Type 1 diabetes, defined as or a HbA1c > 10.0 %, or hospitalization to treat hyper- or hypo-glycemia in the past 3 months within the previous 6 months in participants with Type 2 diabetes
* Participants with severe heart failure, defined as NYHA (New York Heart Association) class IV
* Participants with major surgery including thoracic and cardiac, in the past 3 months, or participants with heart or kidney transplant
* Participants with significant cardiovascular or cerebrovascular events in the past 2 months, such as cardiac arrest, myocardial infarction, or stroke
* Participants with BMI ≥ 40 kg/m2

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2013-02; Primary Completion 2013-07 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Director Clinical Operations, Study Director — Relypsa, Inc.
Locations (58):
- United States (14):
  - Investigator Site 3121, Azusa, California
  - Investigator Site 3133, Los Angeles, California
  - Investigator Site 3103, Sacramento, California
  - Investigator Site 3129, Santa Barbara, California
  - Investigator Site 3130, Ventura, California
  - Investigator Site 3105, Edgewater, Florida
  - Investigator Site 3113, Hollywood, Florida
  - Investigator Site 3106, Port Charlotte, Florida
  - Investigator Site 3120, Augusta, Georgia
  - Investigator Site 3102, Farmington, Missouri
  - Investigator Site 3104, Kansas City, Missouri
  - Investigator Site 3134, Flushing, New York
  - Investigator Site 3107, Bethlehem, Pennsylvania
  - Investigator Site 3110, San Antonio, Texas
- Croatia (5):
  - Investigator Site 1103, Karlovac
  - Investigator Site 1102, Osijek
  - Investigator Site 1104, Zagreb
  - Investigator Site 1105, Zagreb
  - Investigator Site 1106, Zagreb
- Investigator Site 1205, Znojmo, Czechia
- Denmark (4):
  - Investigator Site 2103, Aarhus N
  - Investigator Site 2107, Fredericia
  - Investigator Site 2101, Roskilde
  - Investigator Site 2105, Viborg
- Georgia (12):
  - Investigator Site 1308, Tbilisi
  - Investigator Site 1312, Tbilisi
  - Investigator Site 1301, Tbilisi
  - Investigator Site 1302, Tbilisi
  - Investigator Site 1304, Tbilisi
  - Investigator Site 1305, Tbilisi
  - Investigator Site 1306, Tbilisi
  - Investigator Site 1307, Tbilisi
  - Investigator Site 1309, Tbilisi
  - Investigator Site 1310, Tbilisi
  - Investigator Site 1311, Tbilisi
  - Investigator Site 1303, Tbilisi
- Hungary (7):
  - Investigator Site 1410, Balatonfüred
  - Investigator Site 1415, Budapest
  - Investigator Site 1401, Győr
  - Investigator Site 1406, Hatvan
  - Investigator Site 1405, Jászberény
  - Investigator Site 1411, Kistarcsa
  - Investigator Site 1407, Veszprém
- Investigator Site 2201, Pavia, Italy
- Serbia (3):
  - Investigator Site 1703, Belgrade
  - Investigator Site 1710, Vršac
  - Investigator Site 1707, Zrenjanin
- Slovenia (2):
  - Investigator Site 1802, Celje
  - Investigator Site 1803, Jesenice
- Ukraine (9):
  - Investigator Site 1915, Ivano-Frankivsk
  - Investigator Site 1904, Kharkiv
  - Investigator Site 1903, Kharkiv
  - Investigator Site 1908, Kharkiv
  - Investigator Site 1909, Kyiv
  - Investigator Site 1911, Kyiv
  - Investigator Site 1914, Luhansk
  - Investigator Site 1907, Zaporizhzhia
  - Investigator Site 1906, Zaporizhzhia

REFERENCES:
- [Background] Weir MR, Bakris GL, Bushinsky DA, Mayo MR, Garza D, Stasiv Y, Wittes J, Christ-Schmidt H, Berman L, Pitt B; OPAL-HK Investigators. Patiromer in patients with kidney disease and hyperkalemia receiving RAAS inhibitors. N Engl J Med. 2015 Jan 15;372(3):211-21. doi: 10.1056/NEJMoa1410853. Epub 2014 Nov 21. PMID 25415805
- [Derived] Natale P, Palmer SC, Ruospo M, Saglimbene VM, Strippoli GF. Potassium binders for chronic hyperkalaemia in people with chronic kidney disease. Cochrane Database Syst Rev. 2020 Jun 26;6(6):CD013165. doi: 10.1002/14651858.CD013165.pub2. PMID 32588430

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A Patiromer: Participants were administered patiromer starting dose of 8.4 g or 16.8 g daily as a divided dose twice a day, orally, for 4 weeks.
- Part B Patiromer: Participants continued on the same daily patiromer dose as administered at the time of the Part A Week 4 Visit for 8 weeks.
- Part B Placebo: Participants were administered placebo orally twice a day for 8 weeks.
Period: Part A Treatment Period
Arm/Group | Part A Patiromer | Part B Patiromer | Part B Placebo
Started | 243 | 0 | 0
Completed | 219 | 0 | 0
Not Completed | 24 | 0 | 0
Not completed — Non-compliance with Study Drug | 1 | 0 | 0
Not completed — Protocol Violation | 2 | 0 | 0
Not completed — Adverse Event | 10 | 0 | 0
Not completed — Withdrawal by Subject | 5 | 0 | 0
Not completed — Protocol-specified (eGFR) | 2 | 0 | 0
Not completed — Protocol-specified (High K+) | 3 | 0 | 0
Not completed — Protocol-specified (Low K+) | 1 | 0 | 0
Period: Part B Placebo-Controlled Withdrawal
Arm/Group | Part A Patiromer | Part B Patiromer | Part B Placebo
Started | 0 | 55 (Part A participants with Part A baseline serum potassium ≥ 5.5 mEq/L who responded to treatment) | 52 (Part A participants with Part A baseline serum potassium ≥ 5.5 mEq/L who responded to treatment)
Completed | 0 | 45 | 30
Not Completed | 0 | 10 | 22
Not completed — Physician Decision | 0 | 1 | 1
Not completed — Non-compliance with Study Drug | 0 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 1
Not completed — Death | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Protocol-specified (eGFR) | 0 | 1 | 1
Not completed — Protocol-specified (K+ result) | 0 | 1 | 2
Not completed — Protocol-specified (High K+) | 0 | 2 | 14
Not completed — Protocol-specified (Low K+) | 0 | 2 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Part A Patiromer
Number analyzed (Participants) | 243
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 112
  >=65 years | 131
Age, Continuous [Median (Full Range); unit: years] | 64.2 [29 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103
  Male | 140

OUTCOME MEASURES:

1. Secondary Outcome: Proportion of Participants With Serum Potassium Levels in the Target Range of 3.8 to < 5.1 mEq/L at Part A Week 4
Time Frame: Week 4
Population: Proportion of participants with serum potassium level in the target range at Part A Week 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part A Patiromer
Number analyzed (Participants) | 243
percentage of participants | 76 [70 to 81]
Statistical Analysis 1: Comparison: Part A Patiromer; Test type: Superiority or Other; Proportion = 0.76, 95% CI 2-sided [0.7 to 0.81]

2. Secondary Outcome: Proportion of Participants With Serum Potassium That Was ≥ 5.5 mEq/L in Part B
Time Frame: Part B Baseline to Part B Week 8
Measure: Number; unit: percentage of participants
Arm/Group | Part B Placebo | Part B Patiromer
Number analyzed (Participants) | 52 | 55
percentage of participants | 60 | 15
Statistical Analysis 1: Comparison: Part B Placebo vs Part B Patiromer; Test for difference between treatment groups in proportion with serum potassium ≥ 5.5 mEq/L; Test type: Superiority or Other; p < 0.001, Mantel Haenszel

3. Secondary Outcome: Proportion of Participants With Serum Potassium ≥ 5.1 mEq/L in Part B
Time Frame: Part B Baseline to Part B Week 8
Population: Percentages were estimated not as simple ratios, but by using a stratified method, in order to account for differences between the patiromer and placebo groups in terms of whether participants had type 2 diabetes mellitus and whether they entered the study with serum potassium < 5.8 mEq/L or serum potassium ≥ 5.8 mEq/L.
Measure: Number; unit: percentage of participants
Arm/Group | Part B Placebo | Part B Patiromer
Number analyzed (Participants) | 52 | 55
percentage of participants | 91 | 43
Statistical Analysis 1: Comparison: Part B Placebo vs Part B Patiromer; Test for difference between treatment groups in proportion with serum potassium ≥ 5.1 mEq/L; Test type: Superiority or Other; p < 0.001, Mantel Haenszel

4. Primary Outcome: Change in Serum Potassium From Part A Baseline to Part A Week 4
Description: The primary analysis endpoint is the change from Baseline at Week 4. The estimate of the change at Week 4 is from a repeated measures model, which includes data from Weeks 1, 2, 3 and 4. The analysis includes all intent to treat participants who had a serum potassium result at baseline and at least one weekly post-baseline visit (i.e. Part A Week 1 or later) and excludes six participants who had no result collected after Day 3).
Time Frame: Part A Baseline to Part A Week 4
Measure: Least Squares Mean (Standard Error); unit: mEq/L
Groups:
- Part A Patiromer: Participants were administered patiromer starting dose of 8.4 g or 16.8 g daily as a divided dose twice a day, orally, for 4 weeks. The dose of patiromer could be titrated based on participant's serum potassium response.
Arm/Group | Part A Patiromer
Number analyzed (Participants) | 237
mEq/L | -1.01 (0.031)
Statistical Analysis 1: Comparison: Part A Patiromer; Estimation of mean change in serum potassium from Part A Baseline to Part A Week 4 and test mean change different from zero; Test type: Superiority or Other; p < 0.001, Longitudinal mixed models; Test that the mean change is significantly different from zero

5. Primary Outcome: Change in Serum Potassium From Part B Baseline
Description: Change in Serum Potassium from Part B Baseline to either:
  Part B Week 4 visit, if the participant's serum potassium remained ≥ 3.8 mEq/L and < 5.5 mEq/L up to the Part B Week 4 visit or the earliest Part B visit at which the participant's serum potassium was < 3.8 mEq/L or ≥ 5.5 mEq/L.
Time Frame: Part B Baseline to Part B Week 4 or first local laboratory serum potassium < 3.8 mEq/L or ≥ 5.5 mEq/L
Measure: Median (Inter-Quartile Range); unit: mEq/L
Arm/Group | Part B Placebo | Part B Patiromer
Number analyzed (Participants) | 52 | 55
mEq/L | 0.72 [0.22 to 1.22] | 0 [-0.3 to 0.3]
Statistical Analysis 1: Comparison: Part B Placebo vs Part B Patiromer; Test for difference between treatment groups in serum potassium change in Part B; Test type: Superiority or Other; p < 0.001, ANCOVA

ADVERSE EVENTS:
Time Frame: 2 weeks after Week 4 for Part A subjects who did not continue in Part B and 2 weeks after Week 12 for Part B.
Description: Participants who received at least one dose of trial medication
Arm/Group | Part A Patiromer | Part B Patiromer | Part B Placebo
Serious Adverse Events (participants affected / at risk) | 3/243 | 0/55 | 1/52
Other Adverse Events (participants affected / at risk) | 33/243 | 5/55 | 8/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A Patiromer (N=243) | Part B Patiromer (N=55) | Part B Placebo (N=52)
Anticoagulation drug level below therapeutic (Investigations) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Thrombosis mesenteric vessel (Gastrointestinal disorders) | 0 | 0 | 1
Renal failure chronic (Renal and urinary disorders) | 1 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Endocarditis enterococcal (Infections and infestations) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A Patiromer (N=243) | Part B Patiromer (N=55) | Part B Placebo (N=52)
Hypertension (Vascular disorders) | 4 | 0 | 3
Headache (Nervous system disorders) | 2 | 2 | 4
Constipation (Gastrointestinal disorders) | 26 | 2 | 0
Influenza (Infections and infestations) | 1 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreements generally provide that PI cannot publish single site data before publication of the multi-site publication, unless 1 year has elapsed since completion of the study at all sites. Thereafter, PI may publish provided that PI shall: provide a copy of the publication to sponsor at least 60 days in advance of submission for publication; delete sponsor's confidential information as requested; and delay publication up to an additional 90 days to permit protection of intellectual property.